CLINICAL TRIAL: NCT03684304
Title: The Effect of Abdominal Binder Use on Postoperative Pain and Mobility in Patients Undergoing Pelvic Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Abdominal Binder Use on Postoperative Pain and Mobility in Patients Undergoing Pelvic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients no longer staying overnight in the hospital following this procedure type.
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Caitlin Carlton, Resident Physician, Primary Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: binder071718
Record Dates: First submitted 2018-04-24; First posted 2018-09-25 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Pelvic Organ Prolapse; Abdominal Surgery; Laparoscopic Surgery; Post Operative Pain
MeSH Terms: conditions — Pelvic Organ Prolapse; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control / No Binder (No Intervention): Patients randomized to routine care / no abdominal binder use will not use an abdominal binder during their post operative course.
- Abdominal binder (Experimental): Patients randomized abdominal binder use will have an abdominal binder placed on them in the operating room once their surgery has been completed.
  Interventions: Device: Abdominal binder

INTERVENTIONS:
Device: Abdominal binder — The abdominal binder is an elastic abdominal compression / support device that will be placed on the patient after surgery has been completed.
  Arms: Abdominal binder

SUMMARY:
To determine the effect of post-operative abdominal binder usage on total narcotic usage after undergoing surgery. To determine if abdominal binder usage results in decreased visual analog scale (VAS) pain scores and shorter time to first ambulation post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older.
* Willing and able to provide informed consent.
* Patients must be undergoing scheduled pelvic surgery.
* Patients must be admitted overnight (at least one night) after surgery.

Exclusion Criteria:

* Patients who are younger than 18 years old.
* Patients who are unable or unwilling to provide informed consent.
* Patients who are illiterate.
* Patients who are non-English speaking or reading.
* Patients who are unwilling to be contacted by phone after surgery.
* Patients who are undergoing pelvic surgery that does not warrant observation or admission after surgery for at least one night.
* Patients who are having surgery for any other indication other than pelvic surgery.
* Patients with a chronic pain syndrome (as evidenced by daily intake of opioids).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on female biological sex due to requirement of pelvic surgery.
Enrollment: 36 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control / No Binder | Abdominal Binder
Started | 19 | 17
Completed | 0 | 0
Not Completed | 19 | 17
Not completed — Lost to Follow-up | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control / No Binder | Abdominal Binder | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Full Range); unit: years] | 51 [51 to 51] | 51 [51 to 51] | 51 [51 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: To Assess Effect of Abdominal Binder on Total Post-operative Narcotic Use Within Seven Days Following Pelvic Surgery
Description: Total narcotic usage, calculated in morphine equivalents, during the first seven days post operatively to be calculated and a difference in the amount used by non-abdominal binder patients and abdominal binder patients will be determined. Will review medical record to determine amount of medication used while inpatient, amount / type of narcotic medication prescribed for discharge home, and will call patients to determine how many narcotic pills they have remaining on post operative day seven and calculate the amount used which will then be converted to morphine equivalents.
Time Frame: 7 days
Population: Data not collected
Arm/Group | Control / No Binder | Abdominal Binder
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Assess Whether Post Operative Abdominal Binder Usage Shortens the Time to First Ambulation After Surgery.
Description: Difference in the first time of ambulation after surgery during inpatient admission between non-abdominal binder patients and abdominal binder patients.
Time Frame: 1 day
Population: Data not collected
Arm/Group | Control / No Binder | Abdominal Binder
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Compare Post Operative Pain Scores Using Visual Analog Scale (VAS) Scores in Post Operatives Patients Who Use and do Not Use an Abdominal Binder.
Description: Difference in VAS pain scores will be obtained only while the patient is admitted to the hospital post operatively between non-abdominal binder patients and abdominal binder patients.
Time Frame: 1 day
Population: Data not collected
Arm/Group | Control / No Binder | Abdominal Binder
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Death, serious adverse events, and other were not assessed for this study
Arm/Group | Control / No Binder | Abdominal Binder
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT03684304/Prot_SAP_001.pdf